CLINICAL TRIAL: NCT01115491
Title: A Single Arm Phase II Study of Bevacizumab and Extended Treatment of Temozolomide in Patients With Recurrent Glioblastoma Multiforme
Brief Title: A Study of Bevacizumab and Extended Treatment of Temozolomide in Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25152; 2010-019051-21
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Temozolomide

ARMS (1):
- A (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: temozolomide

INTERVENTIONS:
Drug: bevacizumab [Avastin] — Bevacizumab 10 mg/kg body weight will be administered intravenously every two weeks
Drug: temozolomide — Daily by the oral route (dose, 150 mg/m2) on days 1 to 7 and 15 to 21 of each cycle

SUMMARY:
This is a Phase II, national, multicenter, open-label, non-comparative study to investigate the efficacy and safety of bevacizumab and temozolomide in patients with recurrent glioblastoma multiforme (GBM) after a first treatment failure. Patients will receive bevacizumab 10 mg/kg intravenously every two weeks until disease progression, consent withdrawal, or unacceptable toxicity. Anticipated time on study treatment is 12-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological diagnosis of glioblastoma multiforme (GBM) documented by surgical resection or biopsy.
* They should be patients in a first relapse treated with radiotherapy and chemotherapy and chemotherapy based on temozolomide 150-200 mg/m2 on days 1 to 5 every 28 days (Stupp regimen) for at least three cycles. At least 4 weeks must have lapsed since previous chemotherapy and 3 months since the last dose of radiotherapy.
* Use of an effective contraceptive method by patients and their partners.
* Stable or decreasing corticosteroid dose for the five days prior to study entry
* Adequate hematological function
* Adequate liver function
* Adequate kidney function

Exclusion Criteria:

* Signs of recent bleeding at the MRI of the brain. However, patients with clinically asymptomatic presence of hemosiderin, resolving bleeding changes related to surgery, and presence of punctate hemorrhage in the tumor will be allowed to participate in the study.
* Prior treatment with bevacizumab
* Poorly controlled arterial hypertension
* History of hypertensive crises or hypertensive encephalopathy
* New York Health Association (NYHA) Class II or higher congestive heart failure
* History of myocardial infarction or unstable angina pectoris within six months of study entry
* History of stroke or TIA within six months of study entry
* Significant vascular disease within six months of study entry
* History of hemoptysis > grade 2 according to the NCI CTC criteria within one month of study entry
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgery, open biopsy, intracranial biopsy, ventriculoperitoneal shunt, or major traumatic lesion within 28 days of study entry.
* Core needle biopsy (excluding intracranial biopsy) or other minor surgery within seven days of randomization. Placement of a central vascular access device (CVAD) if performed in the two days prior to bevacizumab administration
* History of abdominal fistula or gastrointestinal perforation within six months of study entry
* History of intracranial abscess within six months of randomization
* Any prior malignant neoplasm treated with curative intent in the five years prior to study entry, except for adequately controlled limited basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix
* Patients with any other metabolic or psychological disease
* Hypersensitivity to products derived from Chinese hamster ovary cells or to other humanized or recombinant human antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Temozolomide: Cycles 1-12 (4-week cycles): Participants received bevacizumab 10 milligrams per kilogram (mg/kg) intravenously (IV) on Days 1 and 15 (followed by 2 weeks off); temozolomide 150 mg per square meter (mg/m^2), orally (PO), on Days 1 through 7 and on Days 15 through 21 (followed by 1 week off). Cycle was repeated for a maximum of 12 cycles.
  Cycle 13 and beyond (4-week cycles): If the first 12 cycles were tolerated with no disease progression, participants then received bevacizumab 10 mg/kg IV on Days 1 and 15 (followed by 2 weeks off). This cycle was repeated every 28 days until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab + Temozolomide
Started | 32
Completed | 2
Not Completed | 30
Not completed — Death | 22
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all enrolled participants.
Groups:
- Bevacizumab + Temozolomide: Cycles 1-12 (4-week cycles): Participants received bevacizumab 10 mg/kg IV on Days 1 and 15 (followed by 2 weeks off); temozolomide 150 mg/m^2, PO, on Days 1 through 7 and on Days 15 through 21 (followed by 1 week off). Cycle was repeated for a maximum of 12 cycles.
  Cycle 13 and beyond (4-week cycles): If the first 12 cycles were tolerated with no disease progression, participants then received bevacizumab 10 mg/kg IV on Days 1 and 15 (followed by 2 weeks off). This cycle was repeated every 28 days until disease progression.
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.19 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time, in weeks, from the date of inclusion in the study to the date of the first documentation of disease progression or death of the participant due to any cause. Participants that did not have an event at the time the analysis was performed were censored at the date of last contact. Participants that began a treatment other than those planned in this study (bevacizumab or temozolomide) were censored on the start date of the new treatment.
Time Frame: Baseline (BL), every 28 days, until progression, death or end-of-study, an average of 32 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
percentage of participants | 96.88

2. Primary Outcome: PFS - Time to Event
Description: PFS was defined as the time, in weeks, from the date of inclusion in the study to the date of the first documentation of disease progression or death of the participant due to any cause. Participants that did not have an event at the time the analysis was performed were censored at the date of last contact. Participants that began a treatment other than those planned in this study (bevacizumab or temozolomide) were censored on the start date of the new treatment. PFS was estimated using the Kaplan-Meier method.
Time Frame: BL, every 28 days, until progression, death or end-of-study, an average of 32 weeks
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
weeks | 18.29 [15.43 to 23.57]

3. Secondary Outcome: Overall Survival - Percentage of Participants With an Event
Description: Overall survival was defined as the time transpired (in weeks) between the date of the participant's inclusion in the trial until the date of his/her death by any cause. Participants that were alive at the time the analysis was performed were censored on the date of last contact.
Time Frame: BL, every 28 days, until death or end-of-study, an average of 32 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
percentage of participants | 75.00

4. Secondary Outcome: Overall Survival - Time to Event
Description: Overall survival was defined as the time transpired (in weeks) between the date of the participant's inclusion in the trial until the date of his/her death by any cause. Participants that were alive at the time the analysis was performed were censored on the date of last contact. Median overall survival was estimated using the Kaplan-Meier method.
Time Frame: BL, every 28 days, until death or end-of-study, an average of 32 weeks
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
weeks | 31.43 [25.14 to 38.29]

5. Primary Outcome: PFS: Probability of Remaining Progression Free at 24 Weeks After Beginning the Study
Time Frame: BL, 24 weeks (after 6th cycle)
Population: ITT population
Measure: Number; unit: survival probability
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
survival probability | 0.30000 (0.0819)

6. Secondary Outcome: Percentage of Participants Achieving an Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Overall response was defined as the percentage of participants who obtained CR or PR using adapted MacDonald criteria. CR: disappearance of all index and non-index lesions, confirmed no less than 4 weeks after assessment, no evidence of disease progression; corticosteroid dosage at or below 20 mg hydrocortisone daily; no neurological changes or an improvement as compared to last disease assessment. PR was defined as: Fifty percent or greater decrease in the sum of products of the larger diameter and the larger perpendicular diameter of all index lesions confirmed no less than 4 weeks after assessment, no evidence of disease progression and the absence of progressive, or non-evaluable disease status for non-index legions; unchanged, or decreased corticosteroid dose as compared to the last disease assessment; no neurological changes or an improvement as compared to the neurological examination at last disease assessment.
Time Frame: BL, every 28 days, until progression, death or end-of-study, an average of 32 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Temozolomide
Number analyzed (Participants) | 32
percentage of participants | 40.6

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the date of start of study treatment to 90 days after the last dose of study treatment.
Description: All participants who received at least 1 dose of study treatment were included in the safety population.
Arm/Group | Bevacizumab + Temozolomide
Serious Adverse Events (participants affected / at risk) | 8/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Temozolomide (N=32)
Lung (pneumonia) (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Fever (General disorders) | 2
Neurological disorder NOS (Nervous system disorders) | 1
Seizures (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 1
Bladder haemorrhage (Renal and urinary disorders) | 1
Intracranial haemorrhage (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Temozolomide (N=32)
Olfactory nerve disorder (Nervous system disorders) | 9
Neurological disorder NOS (Nervous system disorders) | 5
Seizures (Nervous system disorders) | 4
Depressed level of consciousness (Nervous system disorders) | 5
Central nervous system necrosis (Nervous system disorders) | 4
Speech disorder (Nervous system disorders) | 4
Ataxia (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 3
Mood alteration (Nervous system disorders) | 2
Cognitive disturbance (Nervous system disorders) | 2
Lymphocyte count decreased (Blood and lymphatic system disorders) | 16
Platelet count decreased (Blood and lymphatic system disorders) | 15
Neutrophil count decreased (Blood and lymphatic system disorders) | 6
Leukocyte count decreased (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 18
Fever (General disorders) | 4
General symptom (General disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 5
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Upper respiratory infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 2
Lung (pneumonia) (Infections and infestations) | 2
Upper aerodigestive tract infection (Infections and infestations) | 2
Headache (Nervous system disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 7
Glucose, serum-high (hyperglycaemia) (Metabolism and nutrition disorders) | 5
Haemorrhage (General disorders) | 4
Oedema limbs (Blood and lymphatic system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.